CLINICAL TRIAL: NCT06828094
Title: The Effect of Exclusive and Partial Enteral Nutrition on Inflammation-related Proteins and on the Gut Microbiome of Healthy Adults
Brief Title: Enteral Nutrition and Immune Proteins Study
Acronym: ENIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Bernadette White, Miss, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 200220086
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive Enteral Nutrition (Experimental): Replacement of 100% of a participants daily energy intake with enteral nutrition for seven days
  Interventions: Dietary Supplement: enteral nutrition
- Partial Enteral Nutrition (Experimental): Replacement of 50% of a participants daily energy intake with enteral nutrition for seven days
  Interventions: Dietary Supplement: enteral nutrition

INTERVENTIONS:
Dietary Supplement: enteral nutrition — Nutritionally complete liquid diet used in the study to replace all (exclusive enteral nutrition) or half (partial enteral nutrition) of a participants daily energy intake

SUMMARY:
Eligible healthy adults who consent to take part in the study will be randomised to receive either a specialised milkshake for all of their normal daily diet (exculsive enteral nutrition, EEN) or the same specialised milkshake for half of their normal daily diet (partial enteral nutrition, PEN) for seven days. This randomisation is to prevent any bias. In the week before the allocated diet starts participants will be asked to give a weight and height measurement, blood sample, collect a stool and urine sample, and complete a food diary of everything they eat and drink using household measurements (e.g., a teaspoon) seven, four, and one day before the randomly allocated diet begins. Participants will also be asked to give a weight measurement, blood sample, and collect a stool and urine sample before they start the allocated diet. All participants will be asked to collect a third stool, urine, and blood sample and weight measurement at the end of the seven days dietary intervention. Blood samples collected during the study will be used to find out how the cells and proteins which instruct the immune system change during the special milkshake diet. Stool and urine samples will be used to measure the levels of different bacteria which naturally live inside the gut and how their behaviour might have changed during the diet. Those allocated to have PEN will be asked to complete a second set of food diaries for three days during your seven days of specialised milkshake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (>/= 18 years)

Exclusion Criteria:

* Those sufferring from acute or chronic illness (defined as illness which requires regular visits to health services)
* Those who have experienced weight changes +/- 2kg in the past month.
* Previous gut surgery,
* Use of antibiotics or steroids in the past month
* Food allergies which prevent consumption of the enteral nutrition used (milk protein allergy)
* Current pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Changes in Inflammation-Related Proteins | Seven days
  The main outcome measure of this study is to determine changes in inflammation-related proteins in the peripheral blood in response to the seven day dietary intervention.

SECONDARY OUTCOMES:
Changes in Immune Cell Populations | Seven days
  One of the secondary outcome measures is to explore changes in immune cell popultions within the peripheral blood in response to the seven day dietary intervention.
Changes in Gut Microbiome Composition | Seven days
  One of the secondary outcome measures is to explore changes in composition of the gut microbiome in response to the seven day dietary intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided